CLINICAL TRIAL: NCT02272582
Title: A Study to Evaluate the Use of SOMVC001 (GALA) Vascular Conduit Preservation Solution in Patients Undergoing Coronary Artery Bypass Grafting (CABG)
Brief Title: A Study to Evaluate the Use of SOMVC001 (GALA) Vascular Conduit Preservation Solution in Patients Undergoing CABG (STEPS)
Acronym: GALA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Perrault Louis P. (Other)
Collaborators: Montreal Heart Institute (Other); Somahlution LLC (Industry)
Responsible Party: Sponsor-Investigator, Perrault Louis P., Cardiovascular and Thoracic Surgeon, Montreal Heart Institute
Organization: Montreal Heart Institute (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 003-03
Record Dates: First submitted 2014-10-15; First posted 2014-10-23 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOMVC001 Vascular Conduit Solution (Experimental): Each patient will serve as his/her own control because each patient will have two graft segments with one segment immersed in SOMVC001 and the other in heparin dosed saline (Standard solution). Patients will be randomized using a simple random sample allocation scheme. At the time of randomization, patients will be assigned an allocation number. Each randomized patient will be implanted with two SVGs, alternating Target Region A (Circumflex or Diagonal) and Target Region B (Right Coronary System or Diagonal) and alternating (proximal vs. distal) segments of the harvested SV. A randomization schedule will be developed to ensure appropriate randomization allocation of the harvested vein segment being grafted to the targeted regions.
  Interventions: Device: SOMVC001 Vascular Conduit Solution
- Standard of Care Heparin-dosed saline (Active Comparator): Each patient will serve as his/her own control because each patient will have two graft segments with one segment immersed in SOMVC001 and the other in heparin dosed saline (Standard solution). Patients will be randomized using a simple random sample allocation scheme. At the time of randomization, patients will be assigned an allocation number. Each randomized patient will be implanted with two SVGs, alternating Target Region A (Circumflex or Diagonal) and Target Region B (Right Coronary System or Diagonal) and alternating (proximal vs. distal) segments of the harvested SV. A randomization schedule will be developed to ensure appropriate randomization allocation of the harvested vein segment being grafted to the targeted regions.
  Interventions: Other: Standard of care Heparin-dosed saline

INTERVENTIONS:
Device: SOMVC001 Vascular Conduit Solution — SV harvesting will be uniformly performed using an open or endoscopic vein harvesting technique. Once harvested, the SV will be divided into segments and these vein segments from each patient to be immersed in one of two blinded solutions: SOMVC001 or heparin dosed saline. The patients will then be randomized and SVG segment allocations will be defined and grafted to the assigned target regions.
  Arms: SOMVC001 Vascular Conduit Solution
Other: Standard of care Heparin-dosed saline — SV harvesting will be uniformly performed using an open or endoscopic vein harvesting technique. Once harvested, the SV will be divided into segments and these vein segments from each patient to be immersed in one of two blinded solutions: SOMVC001 or heparin dosed saline. The patients will then be randomized and SVG segment allocations will be defined and grafted to the assigned target regions.
  Other Names: active comparator
  Arms: Standard of Care Heparin-dosed saline

SUMMARY:
A prospective randomized, double-blinded, comparative within-person study to evaluate the use of SOMVC001 vs. heparin dosed saline in patients undergoing CABG.

DETAILED DESCRIPTION:
Saphenous vein (SV) harvesting will be performed using an open or endoscopic vein harvesting technique. Once harvested, the SV will be divided into segments and these vein segments from each patient to be immersed in one of two blinded solutions: SOMVC001 or heparin dosed saline. The patients will then be randomized and SVG segment allocations will be defined and grafted to the assigned target regions. Imaging, using 64-slice or better MDCT, will be completed 4-6 weeks and 3 months post surgery (CABG) procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient is to undergo primary, multi-vessel CABG with at least two saphenous vein grafts (SVGs)

Exclusion Criteria:

* Patient has in-situ Internal Mammary Artery graft(s) (IMA) only, (no SVG or free arterial grafts)
* Patients has had prior CABG or planned concomitant valve surgery or aortic aneurysm repair.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-09-24 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
Mean wall thickness of paired grafts within 100 participants measured at 4-6 weeks and 3 months post-CABG surgery using 64-slice multidetector computed tomography (MDCT) angiography. | 4-6 weeks to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Louis P Perrault, MD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Ben Ali W, Voisine P, Olsen PS, Jeanmart H, Noiseux N, Goeken T, Satishchandran V, Cademartiri F, Cutter G, Veerasingam D, Brown C, Emmert MY, Perrault LP. DuraGraft vascular conduit preservation solution in patients undergoing coronary artery bypass grafting: rationale and design of a within-patient randomised multicentre trial. Open Heart. 2018 Apr 13;5(1):e000780. doi: 10.1136/openhrt-2018-000780. eCollection 2018. PMID 29682294